CLINICAL TRIAL: NCT01552564
Title: The Microcirculation in Acute Myocardial Infarction (Micro-AMI)
Acronym: Micro-AMI
Status: Completed | Type: Observational
Sponsor: University of Bristol (Other)
Responsible Party: Principal Investigator, Elisa McAlindon, Clinical Research Fellow, University of Bristol
Other Study IDs: 1625
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- STEMI patients: Consecutive patients presenting through the PPCI service
  Interventions: Procedure: Index of microvascular resistance; Other: Cardiac magnetic resonance; Other: Blood markers

INTERVENTIONS:
Procedure: Index of microvascular resistance
Other: Cardiac magnetic resonance
Other: Blood markers

SUMMARY:
This study investigates the association between the microvascular resistance at the time of primary percutaneous intervention, with microvascular obstruction on CMR and blood markers of myocardial damage.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Cardiac symptoms of > 20 mins chest pain or equivalent.
* ECG criteria consistent with STEMI (STEMI)
* Proceeding with percutaneous angioplasty
* Assent/ consent to the study

Exclusion Criteria:

* Known allergy to adenosine or gadolinium
* Chronic atrial fibrillation
* Renal impairment with eGFR <30
* Contraindication to angiography
* Contraindication to CMR (implanted pacemaker/ defibrillator, ferromagnetic metal implant/ injury, claustrophobia, obesity/ too large for CMR scanner)
* Cardiogenic shock
* Patients with special communication needs or altered consciousness.
* Patients who do not give assent/consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI attending Bristol Heart Institute via the primary PCI service
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Microvascular obstruction | DAy 2-4
  Microvascular obstruction as a percentage of the left ventricle at 2-4 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Bristol Heart Institute, Bristol, United Kingdom

REFERENCES:
- [Derived] McAlindon E, Pufulete M, Harris J, Lawton C, Johnson T, Strange J, Baumbach A, Bucciarelli-Ducci C. Microvascular dysfunction determines infarct characteristics in patients with reperfused ST-segment elevation myocardial infarction: The MICROcirculation in Acute Myocardial Infarction (MICRO-AMI) study. PLoS One. 2018 Nov 13;13(11):e0203750. doi: 10.1371/journal.pone.0203750. eCollection 2018. PMID 30422990